CLINICAL TRIAL: NCT06992882
Title: A Randomized, Open-label, Multi-center Phase III Study Comparing the Efficacy of Oral Chemotherapy Combined With Trastuzumab Versus Paclitaxel Combined With Trastuzumab in the Adjuvant Treatment of HER2-positive, Lymph Node-negative Early Breast Cancer Patients(ORCHID-PLUS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORCHID-PLUS
Record Dates: First submitted 2025-05-20; First posted 2025-05-28 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Capecitabine; Trastuzumab; Paclitaxel

STUDY DESIGN:
Intervention Model Description: In this study, patients who meet the inclusion criteria will be randomized 1:1 to receive capecitabine (1000-1250mg/m2, oral, bid, D1-14, q3w) trastuzumab (first dose 8mg/kg, q3w; Subsequent maintenance 6 mg/kg, q3w, subcutaneous or intravenous for 1 year) or paclitaxel (80 mg/m2, qw, D1, 8, 15, intravenous, q3w) trastuzumab (first dose 8 mg/kg, q3w; Follow-up maintenance 6mg/kg, q3w, subcutaneous or intravenous for 1 year).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XH (Experimental): Capecitabine (1000-1250mg/m2, orally, bid, D1-14, q3w) and trastuzumab (first dose 8mg/kg, q3w; Follow-up maintenance 6 mg/kg, q3w, subcutaneous or intravenous for 1 year)
  Interventions: Drug: Capecitabine
- PH (Experimental): Paclitaxel (80mg/m2, qw, D1, 8, 15, intravenous, q3w) and trastuzumab (first dose 8mg/kg, q3w; Follow-up maintenance 6mg/kg, q3w, subcutaneous or intravenous for 1 year)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Capecitabine — capecitabine (1000-1250mg/m2, orally, bid, D1-14, q3w) and trastuzumab (first dose 8mg/kg, q3w; Follow-up maintenance 6 mg/kg, q3w, subcutaneous or intravenous for 1 year)
  Other Names: Trastuzumab
  Arms: XH
Drug: Paclitaxel — paclitaxel (80mg/m2, qw, D1, 8, 15, intravenous, q3w) trastuzumab (first dose 8mg/kg, q3w; Follow-up maintenance 6mg/kg, q3w, subcutaneous or intravenous for 1 year)
  Other Names: Trastuzumab
  Arms: PH

SUMMARY:
Although there is a certain risk of recurrence of HER2-positive small tumors, the overall prognosis is relatively good. In order to further reduce the toxicity and side effects of treatment and explore the best strategy for adjuvant therapy in patients with HER2-positive stage IA breast cancer, we designed this phase III, randomized, open-label study to evaluate the efficacy and safety of paclitaxel plus trastuzumab and capecitabine versus paclitaxel plus trastuzumab in the adjuvant treatment of patients with HER2-positive, node-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18~70;
2. The postoperative pathological stage of early breast cancer is stage IA: the longest diameter of invasive cancer is not more than 2cm and the lymph node is negative: pT1mic-T1cN0M0 (micro-invasion needs to meet multiple foci).
3. Pathological immunohistochemistry must meet the following conditions: HER-2 (3) or HER-2 (0-2) but amplified by FISH or CISH testing.
4. The maximum number of weeks (56 days) from surgery to randomization is not more than 8 weeks (56 days).
5. The function of major organs is normal, that is, the following criteria are met: (1) The criteria for routine blood examination must meet: HB ≥90 g/L (no blood transfusion within 14 days); ANC ≥1.5×109 /L； PLT ≥100×109 /L； (2) Biochemical tests must meet the following standards: TBIL ≤1.5×ULN (upper limit of normal value); ALT and AST ≤3×ULN; Serum Cr ≤1×ULN, endogenous creatinine clearance >50 ml/min (Cockcroft-Gault formula);
6. Cardiac function: ECG was generally normal, QTc < 470 ms, LVEF >50%;
7. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up

Exclusion Criteria:

1. Patients who have received neoadjuvant therapy, including chemotherapy, targeted, radiotherapy, or endocrine therapy;
2. History of other malignant tumors in the past, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
3. metastasis of any site;
4. Pregnant or lactating women, women of childbearing age who cannot use effective contraception;
5. Patients who are also participating in other clinical trials;
6. Severe organ function (heart, lung, liver, kidney) insufficiency, LEVF < 50% (ultrasound), severe cardiovascular and cerebrovascular diseases (such as: unstable angina, chronic heart failure, uncontrolled hypertension >150/90mmgh, myocardial infarction or cerebrovascular accident) within 6 months before enrollment; Diabetic patients with poor glycemic control; Patients with severe hypertension;
7. Severe or uncontrolled infection;
8. Those who have a history of psychotropic drug abuse and cannot be quit or have a history of mental disorder;
9. Patients who are judged by the investigator to be unsuitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2306 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2028-06-08 (Estimated); Study Completion 2030-06-10 (Estimated)

PRIMARY OUTCOMES:
iDFS | 5 years
  invasive disease-free survival

SECONDARY OUTCOMES:
DDFS | 5 years
  distant disease-free survival
OS | 5 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center Shanghai, China, 200032, Shanghai, Shanghai Municipality, China